CLINICAL TRIAL: NCT01358474
Title: Detecting Dopaminergic Deficits in Individuals At-risk for Parkinsonism
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-DAT-003
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease; Gaucher Disease; Idiopathic Rapid Eye Movement Sleep Disorder
Keywords: Parkinson disease; idiopathic rapid eye movement sleep disorder; Gaucher disease; healthy volunteer
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PD Subjects: Subjects diagnosed with Parkinson's disease (PD)
- At-risk for PD: Subjects at-risk for developing PD (e.g., those with idiopathic rapid eye movement sleep disorder (iRBD) and those who are heterozygous or homozygous for Gaucher's disease (GBA) mutations)
- Healthy Controls: Healthy volunteers

SUMMARY:
The purpose of this study is to determine if participants have changes in dopamine cells in their brain using DaTSCAN™ brain imaging. Dopamine cell loss occurs in Parkinson's disease (PD) and other degenerative Parkinsonian disorders, but does not occur in most other movement disorders such as essential tremor or dystonia. DaTSCAN, which is also known as 123I-Ioflupane, is a new compound that has been developed by General Electric, Inc. and has been approved by the US Food and Drug Administration (FDA) to help doctors detect changes in dopamine. This test is performed by injecting DaTSCAN into a vein in the arm, and after a few hours, a large amount of DaTSCAN temporarily accumulates in an area of the brain where there are a lot of dopamine brain cells. Because DaTSCAN contains a small amount of radioactive iodine, it allows doctors to use a special machine called single photon emission computed tomography (SPECT) scanning to detect the location and amount of radioactivity in the brain and help determine if there are changes in brain dopamine. It is hoped that this study will help doctors detect the presence of dopamine changes even before symptoms are present. This study will evaluate DaTSCAN in people with PD, those who are at risk for developing PD (e.g., those with idiopathic rapid eye movement sleep disorder (iRBD) and those who are heterozygous or homozygous for Gaucher's disease (GBA) mutations) and those who are healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Written consent prior to study by the subject or their surrogate
* Subjects >/= 18 years and</=85 years
* Diagnosis of Parkinson's disease, family history of Parkinson's disease, idiopathic rapid eye movement sleep behavioral disorder, age-matched controls, Gaucher's disease or carrier of Gaucher's gene mutation
* Females using adequate methods of birth control or not of childbearing potential

Exclusion Criteria:

* Any clinically significant acute or unstable physical or psychological disease based on medical history or screening physical examination
* Any exposure to investigational drugs within 4 weeks prior to Visit 1
* Any exposure to radiopharmaceuticals within 4 weeks prior to Visit 1
* Pregnancy
* Breastfeeding
* Severe swallowing problems
* Known sensitivity or allergy to iodine containing products
* Advanced liver or renal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators' clinical practice (e.g., neurology clinic, sleep disorder clinic, etc).
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
single photon computed tomography (SPECT) imaging following administration of a visual adjunct imaging agent that detects dopamine loss | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tuite, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Center for Magnetic Resonance Research, Minneapolis, Minnesota, United States